CLINICAL TRIAL: NCT03830736
Title: Effects of Oat and Oat Components on Cardiometabolic- and Cognitive Test Variables
Brief Title: Health Effects of Oats and Oat Bioactive in Human
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Swedish Foundation for Strategic Research (Other)
Responsible Party: Principal Investigator, Anne Nilsson, Associate professor, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Protokoll 2018/8
Record Dates: First submitted 2019-01-30; First posted 2019-02-05 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Postprandial Glucose Regulation
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: a randomized blinded cross-over study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control product (Placebo Comparator): A glucose solution (glucose and water) based on 42 gram carbohydrates.
  Interventions: Combination Product: Control product
- Oat Beverage 1 (Experimental): The test product is an oat based beverage with added vegetable oil. The test portion is based on 42 gram available carbohydrates and consumed as a breakfast meal prior to determinations of test variables in the morning.
  Interventions: Combination Product: Oat Beverage 1
- Oat Beverage 2 (Experimental): The test product is an oat based beverage with added vegetable oil. The test portion is based on 42 gram available carbohydrates and consumed as a breakfast meal prior to determinations of test variables in the morning.
  Interventions: Combination Product: Oat Beverage 2
- Oat Beverage 3 (Experimental): The test product is an oat based beverage with added vegetable oil. The test portion is based on 42 gram available carbohydrates and consumed as a breakfast meal prior to determinations of test variables in the morning.
  Interventions: Combination Product: Oat Beverage 3
- Oat Beverage 4 (Experimental): The test product is an oat based beverage. The test portion is based on 42 gram available carbohydrates and consumed as a breakfast meal prior to determinations of test variables in the morning.
  Interventions: Combination Product: Oat Beverage 4

INTERVENTIONS:
Combination Product: Oat Beverage 1 — Oat based beverage with added different concentration of extracted oat component.
  Arms: Oat Beverage 1
Combination Product: Oat Beverage 2 — Oat based beverage with added different concentration of extracted oat component.
  Arms: Oat Beverage 2
Combination Product: Oat Beverage 3 — Oat based beverage with added different concentration of extracted oat component.
  Arms: Oat Beverage 3
Combination Product: Oat Beverage 4 — Oat based beverage with added different concentration of extracted oat component.
  Arms: Oat Beverage 4
Combination Product: Control product — Glucose based beverage without added test components is used as control product
  Arms: Control product

SUMMARY:
Aim of the study is to investigate health effects of oats and oat derived components, in human intervention studies, with the purpose to build new knowledge for development of cardiometabolic protective foods.

DETAILED DESCRIPTION:
The overall goal is to increase the knowledge which can be used for the development of food products with anti-diabetic properties, with the purpose to facilitate healthier food choices for people. More specifically the primary purpose of this project is to evaluate effects in healthy humans on cardiometabolic test markers of oat and oat based product. The new knowledge will form a base for the development of oat based food products with added health values.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults
* BMI 18,5 - 25
* non smokers
* consuming a non-vegetarian diet that follows the Nordic guidances

Exclusion Criteria:

* Fasting blood glucose concentration >6.1 mmol/l
* known cardio-metabolic disease (e.g. diabetes, hypertension, metabolic syndrome), gastro-intestinal disorders such as IBS (irritable bowel syndrome) that can interfere with the study results, food allergies. Further no antibiotics or probiotics should have been consumed within 4 weeks prior to and during the study.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Blood glucose regulation | 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Postprandial blood glucose regulation (incremental area under the curve) acute after intake of the test products and at forthcoming meals within 5.5 hours after consumption of test products.

SECONDARY OUTCOMES:
Serum insulin | 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Acute effects of postprandial serum insulin concentrations (incremental area under the curve) after intake of the test products.
plasma GLP-1 (glucagon-like peptide-1 ) | 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Gastro-intestinale hormones involved in appetite and metabolic regulation
IL (interleukin)-6 | 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Inflammatory markers in blood
Plasma PYY (peptide tyrosine tyrosine) | 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Gastro-intestinale hormones involved in appetite and metabolic regulation
IL- 1beta | 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Inflammatory markers in blood

OTHER OUTCOMES:
Subjective appetite sensations | 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Determined with VAS (visual analogue scale) scales (0-100 mm) as a range of subjective sensations related to appetite (such as hunger, desire to eat or fullness)
Breath hydrogen concentrations | 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Indicator of gut fermentation
Mood (valence and activity) | 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Determined with VAS (visual analogue scale) scales 0-100 mm

CONTACTS AND LOCATIONS:
Overall Officials: Anne Nilsson, Study Chair — Lund University
Locations (1):
- Food Technology, engineering and Nutrition, LTH, Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No